CLINICAL TRIAL: NCT04761276
Title: Evaluation of Efficacy and Long-term Safety for Lucidis Instant Focus© - PMCF Study Protocol
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: SAV-IOL SA (Industry)
Collaborators: CEISO (Industry)
Responsible Party: Sponsor
Other Study IDs: LUCIDIS2021
Record Dates: First submitted 2021-02-09; First posted 2021-02-18 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lucidis Intra-ocular lens (IOL): Adult patients with significant reduction in visual acuity and/or visual comfort from cataract who will receive Lucidis Intra-ocular lens
  Interventions: Device: Surgical implantation of intra ocular lens

INTERVENTIONS:
Device: Surgical implantation of intra ocular lens — Cataract surgery may be indicated when the cataract reduces visual function to a level that interferes with everyday activities of the patient leading the patient to desire a surgical intervention to improve its vision.

SUMMARY:
The objectives of the study is to evaluate efficacy and long-term safety of the Lucidis lens. Through this study, the objective is to obtain an up-to-date clinical evaluation of the medical device thus supplementing data from experimental trials. Clinical and functional changes in the implanted eyes among a patient population in which the opaque crystalline lens resulting from cataract was removed and replaced by a Lucidis IOL will be described.

DETAILED DESCRIPTION:
Refractory function in patients with a cataract is mainly restored by implanting intra-ocular lenses (IOL) destined to replace the crystalline lens. While new surgical techniques for removing the crystalline lens have been developed, these lenses have been considerably perfected to resemble the natural crystalline lens as closely as possible.

The objectives of the study is to evaluate efficacy and long-term safety of the Lucidis lens. Through this study, the objective is to obtain an up-to-date clinical evaluation of the medical device thus supplementing data from experimental trials. Clinical and functional changes in the implanted eyes among a patient population in which the opaque crystalline lens resulting from cataract was removed and replaced by a Lucidis IOL will be described.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (≥18 years)
* having agreed to take part in the study and complete post-operative follow-up requirements (by having signed the information leaflet-informed consent form);
* with;
* for whom the physician made the decision to implant a Lucidis

Exclusion Criteria:

* patient included in an interventional therapeutic trial at the time of inclusion;
* patient presenting contraindications for the implantation of an intraocular lens;
* patient presenting an ophthalmic disorder liable to interfere with the study endpoints;
* patient presenting with an astigmatism ≥1.0 D;
* patient refusing or unable to comply with the follow-up procedures in the study (patient unable to be reached by telephone, liable to be lost to follow-up, etc.);
* History of previous intraocular surgery in the study eye in the previous 6 months;
* patient is pregnant, breast-feeding or unable to make the decision to participate in a clinical investigation (e.g. mentally ill or handicapped person)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with significant reduction in visual acuity and/or visual comfort from cataract requiring intra ocular lens implantation
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-05-21 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Visual acuity measure BCVA photopic | 1 year
  Far Best Corrected Visual Acuity in photopic conditions
Visual acuity measure UCVA photopic | 1 year
  Near, intermediate and far Uncorrected visual acuity in photopic conditions
Visual acuity measure BCVA mesopic | 1 year
  Far Best Corrected Visual Acuity in mesopic conditions
Visual acuity measure UCVA mesopic | 1 year
  Near, intermediate and far Uncorrected visual acuity in mesopic conditions

SECONDARY OUTCOMES:
Contrast sensitivity measure photopic | 1 year
  Contrast sensitivity in photopic conditions
Contrast sensitivity measure mesopic | 1 year
  Contrast sensitivity in mesopic conditions
Safety assessment | 1 year
  Adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: Kate Hashemi, Pr, Principal Investigator — Institut jules gonin
Locations (1):
- Hôpital Jules Gonin, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: SAV IOL website — https://sav-iol.com/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/76/NCT04761276/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/76/NCT04761276/ICF_001.pdf